CLINICAL TRIAL: NCT00748319
Title: Analysis of Killer Immunoglobulin-like Receptor Transcripts Expression for the Diagnosis of Epidermotropic Cutaneous T-cell Lymphomas (Mycosis Fungoid and Sézary Syndrome) in Patients With Erythroderma or Erythematous Patches/Plaques.
Brief Title: Killer Immunoglobulin-Like Receptor Transcripts Expression for the Diagnosis of Epidermotropic Cutaneous T Cell Lymphoma
Acronym: KIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070153
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Mycosis Fungicides; Sezary Syndrome; Dermatitis; Dermatitis, Exfoliative
Keywords: Receptors KIR; Polymerase chain reaction; Diagnosis; Lymphoma T-cell cutaneous; Mycosis fungicides; Sezary syndrome; Differential diagnosis from dermatitis
MeSH Terms: conditions — Sezary Syndrome; Dermatitis; Dermatitis, Exfoliative; Disease; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Detection of KIR receptor
  Interventions: Other: Detection of KIR receptor by RT PCR

INTERVENTIONS:
Other: Detection of KIR receptor by RT PCR — Detection on biopsy cutaneous (3mm) and on blood sample of 30 ml

SUMMARY:
The most frequent cutaneous T-cell lymphomas (CTCL) are mycosis fungoid and Sezary syndrome. The diagnosis of these lymphomas is difficult using current methods, especially because numerous benign dermatological conditions can mimick CTCL both clinically and under microscopic examination. Recently, the KIR receptor CD158k has been shown to be a marker for Sezary syndrome in both the blood and skin. We hypothesize that other receptors from the same family may help fro the diagnosis of these lymphomas. To address this issue, we will study the expression of all known KIR receptor in the skin of patients presenting with a skin eruption, which may correspond to either a cutaneous T-cell lymphoma or a benign dermatological disease. The final diagnosis will be established by a panel of experts, allowing constitution of 2 groups of patients : the cutaneous T-cell lymphoma group, and the benign inflammatory disease group. The expression of the different KIRs will be analyzed in both group in a blinded fashion, in order to determine whether one or a several KIRs may be differentially expressed.

DETAILED DESCRIPTION:
Background : The most frequent cutaneous T-cell lymphomas (CTCL) are mycosis fungoid and Sezary syndrome. Both are due to the proliferation of a CD4+ T-cell clone in the skin, associated with a blood involvement in Sezary syndrome. Mycosis fungoid clinically presents as a patches or plaques dermatitis and Sezary syndrome as an exfoliative dermatitis. The diagnosis of these lymphomas is difficult using current methods, especially because numerous benign dermatological inflammatory conditions can mimick CTCL both clinically and under microscopic examination. Recently, the KIR receptor CD158k has been shown to be a marker for Sezary syndrome in both the blood and skin. We hypothesize that other receptors from the same family may help fro the diagnosis of these lymphomas.

Aim of the study : to determine if one or a panel of KIR(s) receptor(s) may help for the differential diagnosis between cutaneous T-cell lymphoma (CTCL) and benign inflammatory dermatoses.

Subjects selection : all patients presenting to an investigator, member of the GFELC experts group ("French Group Study Cutaneous Lymphoma"), with either an exfoliative or patch/plaque dermatitis with a clinical suspicion of CTCL will be enrolled.

Number of subjects : A total of 550 patients could be recruited by the GFELC, including 180 CTCL (60 Sezary syndrome and 120 mycosis fungoid) and 370 inflammatory diseases (240 patch dermatitis and 130 exfoliative dermatitis).

Inclusion period : patients will be included during a 2 years period and will be followed during 6 months. Total study length will be 30 months.

Interventions : 1) 3 mm punch skin biopsy for all patients 2) 10 ml blood sample for patients with exfoliative dermatitis Methods : Following initial and 6 month follow-up evaluations, patients will be classified in one of the following groups : the cutaneous T-cell lymphoma group, and the benign inflammatory disease group. The expression of all known KIRs receptors (KIR2DL1 (CD158a), KIR2DL2 (CD158b1), KIR2DL3 (CD158b2), KIR2DL4 (CD158d), KIR2DL5 (CD158f), KIR3DL1 (CD158e1), KIR3DL2 (CD158k), KIR2DS1 (CD158h), KIR2DS2 (CD158j), KIR2DS4 (CD158i), KIR2DS5 (CD158g), KIR3DS1 (CD158e2)) will be evaluated using reverse transcription and quantitative polymerase chain reaction in all skin and blood samples, in a blinded fashion. For blood samples, the analyses will be performed on CD4+ T-cell sorted using magnetic beads.

Outcome measures : The main outcome measure will be the differential expression of one or a panel of KIR(s) receptor(s) between CTCL and benign inflammatory diseases. Secondary outcome measure will be a differential quantitative expression of one or a panel of KIR(s) receptor(s) between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Subacute/chronic dermatitis (>7 days) with clinical suspicion for cutaneous T-cell lymphoma
* No past history of lymphoma or other hematologic malignancy
* Skin biopsy for routine histology at inclusion
* Cutaneous T-cell clonality analysis at inclusion
* Sezary cell count on routine blood smear examination in case of erythroderma
* Blood T-cell clonality analysis at inclusion in case of erythroderma
* Age<18 years
* Skin biopsy for routine histology at inclusion (Possibility, in the 6 previous months of inclusion without any specific treatment other taht local corticoids- amendment n°4)
* Cutaneous T-cell clonality analysis at inclusion (Possibility, in the 6 previous months of inclusion without any specific treatment other taht local corticoids- amendment n°4)
* Realization of a preliminary medical examination
* Sezary cell count on routine blood smear examination in case of erythroderma (Possibility, in the 6 previous months of inclusion without any specific treatment other taht local corticoids- amendment n°4)
* Blood T-cell clonality analysis at inclusion in case of erythroderma (Possibility, in the 6 previous months of inclusion without any specific treatment other taht local corticoids- amendment n°4)

Exclusion Criteria:

* Adults under tutelage
* Subject not affiliated at the French National health and pensions organization

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Differential expression of one or a panel of KIRs transcript(s) between epidermotropic cutaneous lymphoma and inflammatory diseases | at the inclusion

SECONDARY OUTCOMES:
Difference(s) in the quantitative expression of one or a panel of KIRs transcript(s) between epidermotropic cutaneous lymphoma and inflammatory diseases | at the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Ortonne, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe hospitalier Henri Mondor - Albert Chenevier, Créteil, France